CLINICAL TRIAL: NCT04488783
Title: Potentiation of Chemotherapy in Brain Tumors by Zinc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Leor Zach, MD, MD, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4266-17-SMC
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Newly Diagnosed Glioblastoma Who Underwent at Least Partial Resection of the Tumor Surgically
Keywords: GBM; glioblastoma; zinc; vitamin C
MeSH Terms: conditions — Glioblastoma | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glioblastoma patients (Experimental): newly diagnosed GB who underwent at least partial resection of the tumor surgically
  Interventions: Dietary Supplement: zinc and ascorbate

INTERVENTIONS:
Dietary Supplement: zinc and ascorbate — oral zinc and ascorbate

SUMMARY:
Glioblastoma (GB) is the most common and aggressive type of primary malignant brain tumor in adults. Despite advances in surgical resection, radiotherapy and chemotherapy, prognosis remains very poor. Temozolomide (TMZ) as an alkylating agent has become part of GBM management but it has contributed only marginally to prolongation of life in GBM patients. Our aim is to evaluate the therapeutic potential of the trace element zinc to facilitate temozolomide tumor cell toxicity in GBM. P53 gene is inactive/mutant in most of these patients which may affect the resistance to apoptosis of tumor cells by chemotherapy. Zinc (Zn) has a crucial role in the biology of p53, in that p53 binds to DNA through a structurally complex domain stabilized by zinc atom. We have shown that the cytotoxic activity of TMZ is substantially increased with the addition of zinc in vitro with GBM cell lines as well as in vivo, with intracranial GBM xenografts. Numerous studies of zinc in animal models and in human subjects support its use in the treatment and possibly the prevention of cancer. Zinc has been consumed by the public as an essential mineral (and thus is category A drug) in concentrations which allows this effect with Temozolomide. Vitamin C could add to this by priming the immune system for lymphocyte- linked cancer killing. The vitamin c increases the number of tumor infiltrating lymphocytes and enhances the activation of the immune system.We propose a single arm phase II clinical trial in 30 newly diagnosed GBM patients who will be treated with the standard chemo-radiotherapy with the addition of zinc and vitamin C.

DETAILED DESCRIPTION:
We propose a single arm phase II clinical trial in 30 newly diagnosed GBM patients who will be treated with the standard chemo-radiotherapy with the addition of daily zinc. We will follow the toxicity, Progression free survival and overall survival of this group of patients. We hope to demonstrate the anti-tumor activity of zinc that will enhance the activity of temozolomide chemotherapy in adult glioblastoma patients. We will also follow the safety and monitor quality of life during treatment. In this study, we will compare results of patients receiving zinc to historical patient data. We will review patient portfolios with GB tumors that received treatment as the subjects in this study in the last five years before the study began. Collecting the data and separating the identified data from the file in a way that cannot be retrieved in any way will be done by a staff member from Dr Ruty Shai's laboratory who is authorized to open medical files. We will adjust the age and number of patients in each gender. Data collected: date of birth, age of disease development, gender, data after receiving treatment: Progression free survival and overall survival of this group of patients, side effects, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females,
* age ≥ 18 years old,
* newly diagnosed GBM, Karnofsky performance status of ≥ 70,
* after partial resection or gross tumor resection (GTR) who recovered from surgical resection.

Exclusion Criteria:

* GB patients with less than 20% of tumor removed,
* Prior treatment for GB (other than surgical resection),
* any known malignancy outside of the brain in the last 5 years,
* in ability to swallow drugs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | year 1
overall survival (OS) | year 2

SECONDARY OUTCOMES:
Tcell count | year 2
  Blood test
Level of Interleukin 6 | year 2
  Interleukin 6 and Tumor Necrosis Factor quantification
Tumor Necrosis Factor quantification | year 2
  Blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No